CLINICAL TRIAL: NCT04485650
Title: The Effect of Music Therapy on Postoperative Pain Anxiety and Vital Signs in Patients Undergoing Spinal Anaesthesia: a Randomized Controlled Trial
Brief Title: Effect of Music in Intraoperative Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: AIBU-AML-UY-01
Record Dates: First submitted 2020-04-24; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Music Therapy; Perioperative Care; Postoperative Pain; Anxiety; Total Knee Arthroplasty; Vital Signs; Spinal Anesthesia
Keywords: music therapy; perioperative care; postoperative pain; anxiety; total knee arthroplasty; vital signs; spinal aesthesia
MeSH Terms: conditions — Pain, Postoperative; Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: In the study, 30 patients were assigned to the music group, 30 patients were assigned to the group that received sedation and 30 patients were assigned to a group that was not sedated, all occurred in a randomized controlled way.
  The music were chosen by a researcher under guidance of an expert and grouped as relaxing, classical, mystical, and Turkish folk music. One of them was chosen by the patients following the application of spinal anesthesia in the music group. Sedation (Dormicum) was performed to the sedated group after spinal anesthesia based on the height and weight data and the doctor's decision. The patients in the non-sedated group were followed without any procedure (sedation and music).
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music group (Experimental): The music were chosen by a researcher under guidance of an expert and grouped as relaxing, classical, mystical, and Turkish folk music. One of them was chosen by the patients following the application of spinal anesthesia in the music group. The number of participants:30
  Interventions: Other: music therapy
- Sedated group (Active Comparator): Sedation was performed to the sedated group after spinal anesthesia based on the height and weight data and the doctor's decision. The number of participants:30
  Interventions: Other: sedated group
- Non-sedated group (Other): The patients in the non-sedated group were followed without any procedure (sedation and music). The number of participants:30
  Interventions: Other: non-sedated group

INTERVENTIONS:
Other: music therapy — The music were chosen by a researcher under guidance of an expert and grouped as relaxing, classical, mystical, and Turkish folk music. One of them was chosen by the patients following the application of spinal anesthesia in the music group.
  Arms: Music group
Other: sedated group — Sedation was performed to the sedated group after spinal anesthesia based on the height and weight data and the doctor's decision. The number of participants:30
  Arms: Sedated group
Other: non-sedated group — The patients in the non-sedated group were followed without any procedure (sedation and music). The number of participants:30
  Arms: Non-sedated group

SUMMARY:
Background and Aims: Music therapy has a wide range of uses in health care practice. The aim of this study was to investigate the effects of intraoperative music played during spinal anesthesia operation on the patients' intraoperative vital signs, postoperative pain, and anxiety status.

Methods: The study was performed in an operating room with a total of 90 patients, of whom 30 were in the music group, 30 were in the control group and 30 were in the sedated group. The ethics committee's approval, institutional permission, and the study participants' written informed consent were obtained. Data were collected using patient information and intraoperative observation form for vital signs as well as through the Visual Analog Scale and State Anxiety Scale. Preoperative and postoperative anxiety, the intraoperative and postoperative vital signs and postoperative pain and anxiety of all groups were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* The patients that had an orthopedic operation
* The patients who took spinal anesthesia
* able to understand, read and speak Turkish, so they may complete the informed consent and questionaires
* Aged 18 or older
* Have a Body Mass Index (BMI) <40
* ASA (American Society of Anaesthesiologists) I-II-III statuses.

Exclusion Criteria:

* Patients with vision and hearing problems and inability to complete questionnaires,
* The patients not have psychiatric disease history and psychiatric drug use,
* The patients not have diseases that could be evaluated as severe (such as heart, kidney, liver failure)
* The patients not underwent emergency surgeries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2017-03-15 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Distribution of systolic blood pressure of patients in the sedated, music and control groups in intraoperative and postoperative period follow-ups | Change from Baseline Systolic Blood Pressure on intraoperative 5 minutes to 2 hours ; postoperative 10 minutes to 2 hours postoperative
  Measurement of systolic blood pressure of patients in the sedated, music and control groups in intraoperative and postoperative period follow-ups
Distribution of diastolic blood pressure of patients in the sedated, music and control groups in intraoperative and postoperative period follow-ups | Change from Baselinebdiastolic Blood Pressure on intraoperative 5 minutes to 2 hours ; postoperative 10 minutes to 2 hours postoperative
  Measurement of diastolic blood pressure of patients in the sedated, music and control groups in intraoperative and postoperative period follow-ups
Distribution of pulse rates of patients in the sedated, music and control groups in intraoperative and postoperative period follow-ups | Change from Baseline pulse rates on intraoperative 5 minutes to 2 hours ; postoperative 10 minutes to 2 hours postoperative
  Measurement of pulse rates of patients in the sedated, music and control groups in intraoperative and postoperative period follow-ups
Distribution of respiratory rates of patients in the sedated, music and control groups in intraoperative and postoperative period follow-ups | Change from Baseline of patients respiratory rates on intraoperative 5 minutes to 2 hours ; postoperative 10 minutes to 2 hours postoperative
  Measurement of respiratory rates of patients in the sedated, music and control groups in intraoperative and postoperative period follow-ups
anxiety assessment 30 minutes before surgery | State- Trait Anxiety Scale was applied to all three groups in 30 minutes before surgery
  State- Trait Anxiety Scale was applied to all three groups in preoperative period.Distribution of preoperative and postoperative state anxiety scores according to groups. State- Trait Anxiety Scale: This scale was developed by Spielberger et al. in 1970 to determine the level of the individual anxiety state. It has 40 items in two constructs of state and trait. Since state anxiety scale was emphasized in the present study, only 20-item state scale construct was used. Each item had a 4-point Likert scale answer, from 1 (almost never) to 4 (almost always), and the possible total score ranged from 20 (the lowest level of anxiety) to 80 (the highest level of anxiety)
anxiety assessment 8 hours after surgery | State- Trait Anxiety Scale was applied to all three groups in 8 hours after surgery
  State- Trait Anxiety Scale was applied to all three groups in postoperative period.Distribution of preoperative and postoperative state anxiety scores according to groups. State- Trait Anxiety Scale: This scale was developed by Spielberger et al. in 1970 to determine the level of the individual anxiety state. It has 40 items in two constructs of state and trait. Since state anxiety scale was emphasized in the present study, only 20-item state scale construct was used. Each item had a 4-point Likert scale answer, from 1 (almost never) to 4 (almost always), and the possible total score ranged from 20 (the lowest level of anxiety) to 80 (the highest level of anxiety)
pain assessment in the operating room | The pain was assessed at the end of the operation in 10 minutes with numerical pain scale
  The pain was assessed with numerical pain scale. Numerical Pain Scale: It is used by the patient himself/herself to assess and measure severity of the pain. The scale begins with the absence of pain (0) and ends at the level of unbearable pain
Postoperative pain at 1 hours | The pain was assessed followed at 1 hours postoperative period with numerical pain scale
  The pain was assessed with numerical pain scale. Numerical Pain Scale: It is used by the patient himself/herself to assess and measure severity of the pain. The scale begins with the absence of pain (0) and ends at the level of unbearable pain.
Postoperative pain at 8 hours | The pain was assessed followed at 8 hours postoperative period with numerical pain scale
  The pain was assessed with numerical pain. Numerical Pain Scale: It is used by the patient himself/herself to assess and measure severity of the pain. The scale begins with the absence of pain (0)

CONTACTS AND LOCATIONS:
Overall Officials: ümmühan yiğit, msc, Principal Investigator — research assistant; arzu ilçe, proffesor, Principal Investigator — faculty of health science of dean; ibrahim karagöz, phd, Principal Investigator — anesthesiology and reanimation doctor
Locations (1):
- Faculty of health sciences, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
when the planned number of participants was reached, the data were coded in a statistical program and shared with other researchers

REFERENCES:
- [Background] Koc H, Erk G, Apaydin Y, Horasanli E, Yigitbasi B, Dikmen B. The Effects of Classical Turkish Music on Patients Undergoing Inguinal Hernia Repair under Epidural Anesthesia. Turk Anaesth Int Care. 2009;37:366-373.
- [Background] Sener EB, Koylu N, Ustun FE, Kocamanoglu S, Ozkan F. The effects of music, white noise and operating room noise on perioperative anxiety in patients under spinal anesthesia. European Journal Of Anaesthesiology (EJA). 2010;24:133
- [Background] Uyar M, Akin Korhan E. [The effect of music therapy on pain and anxiety in intensive care patients]. Agri. 2011 Oct;23(4):139-46. doi: 10.5505/agri.2011.94695. Turkish. PMID 22290677
- [Background] Bansal P, Kharrod U, Sanwatsarkar S, Patel H, Kamat H. The Effect Of Music Therapy On Sedative Requirements And Haemodynamic Parameters In Patients Under Spinal Anaesthesia; A Prospective Study. Journal Of Clinical And Diagnostic Research. 2010;4:2782-2789.
- [Background] Liu Y, Petrini MA. Effects of music therapy on pain, anxiety, and vital signs in patients after thoracic surgery. Complement Ther Med. 2015 Oct;23(5):714-8. doi: 10.1016/j.ctim.2015.08.002. Epub 2015 Aug 4. PMID 26365452
- [Background] Allen K, Golden LH, Izzo JL Jr, Ching MI, Forrest A, Niles CR, Niswander PR, Barlow JC. Normalization of hypertensive responses during ambulatory surgical stress by perioperative music. Psychosom Med. 2001 May-Jun;63(3):487-92. doi: 10.1097/00006842-200105000-00019. PMID 11382277
- [Background] Bae I, Lim HM, Hur MH, Lee M. Intra-operative music listening for anxiety, the BIS index, and the vital signs of patients undergoing regional anesthesia. Complement Ther Med. 2014 Apr;22(2):251-7. doi: 10.1016/j.ctim.2014.02.002. Epub 2014 Feb 23. PMID 24731896
- [Background] Komurcu E, Kiraz HA, Kaymaz B, Golge UH, Nusran G, Goksel F, Sahin H, Omur D, Hanci V. The effect of intraoperative sounds of saw and hammer on psychological condition in patients with total knee arthroplasty: prospective randomized study. ScientificWorldJournal. 2015;2015:690569. doi: 10.1155/2015/690569. Epub 2015 Feb 22. PMID 25793222
- [Background] Sarkar D, Chakraborty K, Bhadra B, Ghorai TK, Singh R, Mandal U. Effects of music on patients undergoing orthopaedic surgery under spinal anaesthesia. IOSR Journal of Dental and Medical Sciences. 2015;14:2279-2861.
- [Background] Chou MH, Lin MF. Exploring the listening experiences during guided imagery and music therapy of outpatients with depression. J Nurs Res. 2006 Jun;14(2):93-102. doi: 10.1097/01.jnr.0000387567.41941.14. PMID 16741859
- [Background] Bailey L. Strategies for decreasing patient anxiety in the perioperative setting. AORN J. 2010 Oct;92(4):445-57; quiz 458-60. doi: 10.1016/j.aorn.2010.04.017. PMID 20888947
- [Background] Boker A, Brownell L, Donen N. The Amsterdam preoperative anxiety and information scale provides a simple and reliable measure of preoperative anxiety. Can J Anaesth. 2002 Oct;49(8):792-8. doi: 10.1007/BF03017410. PMID 12374706
- [Background] Carr E, Brockbank K, Allen S, Strike P. Patterns and frequency of anxiety in women undergoing gynaecological surgery. J Clin Nurs. 2006 Mar;15(3):341-52. doi: 10.1111/j.1365-2702.2006.01285.x. PMID 16466484
- [Background] Gursoy A A. Anxiety Levels of Preoperative Patients and Determining the Factors That May Cause Anxiety. Journal of Nursing Research. 2001;1:23-29.
- [Background] Turhan Y, Avci R, Ozcengiz D. The Relationship Between Preoperative And Postoperative Anxiety, And Patient Satisfaction In Preparation For Elective Surgery. Journal of Anesthesia. 2012;20:27-33
- [Background] Vaughn F, Wichowski H, Bosworth G. Does preoperative anxiety level predict postoperative pain? AORN J. 2007 Mar;85(3):589-604. doi: 10.1016/S0001-2092(07)60130-6. PMID 17352896
- [Background] Yilmaz E, Aydin E. The Effect of Pre and Postoperative Anxiety in Quality of Recovery in Patients Undergoing Surgery. Fırat Health Services Journal. 2013;8:79-95.
- [Background] Eti Aslan F. The assessment methods of pain. Journal of Cumhuriyet University School of Nursing. 2002;6:9-16.
- [Background] Shek DT. The Chinese version of the State-Trait Anxiety Inventory: its relationship to different measures of psychological well-being. J Clin Psychol. 1993 May;49(3):349-58. doi: 10.1002/1097-4679(199305)49:33.0.co;2-j. PMID 8315037
- [Background] Lepage C, Drolet P, Girard M, Grenier Y, DeGagne R. Music decreases sedative requirements during spinal anesthesia. Anesth Analg. 2001 Oct;93(4):912-6. doi: 10.1097/00000539-200110000-00022. PMID 11574356
- [Background] Zhu NN, Xu PP, Lei TT, Sun T, Chan SW. Postoperative Pain Self-Management Behavior in Patients Who Underwent Total Knee or Hip Arthroplasty. AORN J. 2017 Apr;105(4):355-364. doi: 10.1016/j.aorn.2017.02.001. PMID 28336024
- [Background] Chen HJ, Chen TY, Huang CY, Hsieh YM, Lai HL. Effects of music on psychophysiological responses and opioid dosage in patients undergoing total knee replacement surgery. Jpn J Nurs Sci. 2015 Oct;12(4):309-19. doi: 10.1111/jjns.12070. Epub 2015 Mar 9. PMID 25754254
- [Background] Sendelbach SE, Halm MA, Doran KA, Miller EH, Gaillard P. Effects of music therapy on physiological and psychological outcomes for patients undergoing cardiac surgery. J Cardiovasc Nurs. 2006 May-Jun;21(3):194-200. doi: 10.1097/00005082-200605000-00007. PMID 16699359
- [Background] Ozdemir U, Tasci S, Yildizhan E, Aslan S, Eser B. The Effect of Classical Turkish Music on Pain Severity and Anxiety Levels in Patients Undergoing Bone Marrow Aspiration and Biopsy. Pain Manag Nurs. 2019 Feb;20(1):82-87. doi: 10.1016/j.pmn.2018.04.009. Epub 2018 May 18. PMID 29784556
- [Background] Labrague LJ, McEnroe-Petitte DM. Influence of Music on Preoperative Anxiety and Physiologic Parameters in Women Undergoing Gynecologic Surgery. Clin Nurs Res. 2016 Apr;25(2):157-73. doi: 10.1177/1054773814544168. Epub 2014 Jul 30. PMID 25078946
- [Background] Jimenez-Jimenez M, Garcia-Escalona A, Martin-Lopez A, De Vera-Vera R, De Haro J. Intraoperative stress and anxiety reduction with music therapy: a controlled randomized clinical trial of efficacy and safety. J Vasc Nurs. 2013 Sep;31(3):101-6. doi: 10.1016/j.jvn.2012.10.002. PMID 23953858

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-20): https://cdn.clinicaltrials.gov/large-docs/50/NCT04485650/Prot_SAP_000.pdf